CLINICAL TRIAL: NCT03412188
Title: Evaluation of the Effect of Eltrombopag on the Expression of Platelet Collagen Receptor Glycoprotein VI (GPVI) in Pediatric Patients With Chronic and Persistent Immune Thrombocytopenia.
Brief Title: The Effect of Eltrombopag on the Expression of Platelet Collagen Receptor GPVI in Pediatric ITP.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nayera Hazaa Elsherif (Other)
Responsible Party: Sponsor-Investigator, Nayera Hazaa Elsherif, assistant professor of pediatrics, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GPVI-ITP
Record Dates: First submitted 2018-01-20; First posted 2018-01-26 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Idiopathic Thrombocytopenic Purpura
Keywords: Chronic ITP; persistent ITP; Eltrombopag; GPVI receptor
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag; Congresses as Topic; Methylprednisolone Hemisuccinate; Azathioprine; Mycophenolic Acid; Rituximab

STUDY DESIGN:
Intervention Model Description: Patients will be divided into 2 groups:
  Group 1 (eltrombopag arm n=20 patients): Patients who showed no response (platelet count ≤ 20x109/L) initially for 3 months or relapse after 6 months after at least one prior ITP therapy. patients will receive a total daily dose of eltrombopag of (25-50mg/d). Dose adjustments may be made based on platelets count.
  Group 2 (n=20 patients) Patients who are currently receiving other lines of treatment (steroids, IVIG, azathioprine, and rituximab).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1 Eltrombopag arm (Experimental): Group 1 (eltrombopag arm n=20 patients): Patients who showed no response (platelet count ≤ 20x109/L) initially for 3 months or relapse after 6 months after at least one prior ITP therapy. patients will receive a total daily dose of eltrombopag of (25-50mg/d). Dose adjustments may be made based on platelets count with an increment of 25mg once per day at 2 weeks intervals (Maximum dose: 75 mg orally once a day).
  Patients, who responded poorly to eltrombopag in 6 months or developed adverse effects, were asked to discontinue the medication. Those who responded were followed for further 6 month period.
  Interventions: Drug: Eltrombopag
- group 2 conventional Treatment (Active Comparator): Group 2 (n=20 patients) Patients who are currently receiving other lines of treatment (steroids, IVIG, azathioprine, and rituximab).
  patients will continue on the conventional line of treatment
  Interventions: Drug: conventional

INTERVENTIONS:
Drug: Eltrombopag — Patients who showed no response (platelet count ≤ 20x109/L) initially for 3 months or relapse after 6 months after at least one prior ITP therapy will receive a total daily dose of eltrombopag of (25-50mg/d)
  Other Names: Revolade
  Arms: group 1 Eltrombopag arm
Drug: conventional — Patients who are currently receiving conventional lines of treatment (steroids, IVIG, azathioprine, and rituximab, Mycophenolate mofetil) will continue on the same line of treatment
  Other Names: solumedrol; imuran; cellcept; mabthera; gammaglobulin
  Arms: group 2 conventional Treatment

SUMMARY:
Using eltronmobag as an alternative pathway, which depend on stimulation of thrombocyte synthesis, in chronic and persistent immune thrombocytopenia may be more promising treatment than the classic type, not only by increasing platelets count but also through enhancing of the platelets activation and upregulation of GPVI expression on platelet surface.

This study will include 40 pediatric patients with chronic or persistent ITP, recruited from the Hematology clinic of pediatric hospital Ain Shams University, aiming to investigate the efficacy, & the safety and tolerability of eltrombopag therapy for children as well as the ability of eltrombopag to enhance the platelet activation through the up-regulation of glycoprotein VI (GPVI) receptor expression in comparison with other lines of treatment.

Patients will be divided into 2 groups : Group 1 on eltrombopag ; Group 2 : receiving other lines of therapy .

All Patients will be subjected to :

1. bleeding score assessment ( baseline &every month ) and Health related quality of life based on Kids' ITP Tools (KIT) questionnaires( baseline and week 24 )
2. Baseline and at week 24 bone marrow examination with reticulin stain
3. clinical examination every 2 weeks and complete blood counts.
4. Assessment of soluble form of glycoprotein VI using sandwich enzyme-linked immunosorbent assay (ELISA) as well as assessment of platelet activation by GPVI using flowcytometry (Gardiner, etal.,2010 ) at baseline and at the end of 6 months treatment period

DETAILED DESCRIPTION:
Primary immune thrombocytopenia (ITP) is an acquired immune-mediated disorder characterized by isolated thrombocytopenia, defined as a peripheral blood platelet count less than 100 ×109/l and the absence of any obvious initiating and/ or underlying cause of the thrombocytopenia. (Buchanan, 1989).

Novel thrombopoiesis-stimulating agents have been developed increasing platelet production by overdriving the system and thereby correcting the thrombocytopenia (Cines etal., 2002). Because these peptides bear no structural resemblance to thrombopoietin agonist(TPO) but still bind and activate the TPO receptor, these compounds are called TPO receptor agonists (TRAs). (Meletis etal.,2010).

Newly formed young platelets are larger and express higher levels of glycoprotein Ibα (GPIbα), which decreases as platelets age. For the purpose of quantitative platelet analysis, GPIbα of the GPIb-IX-V complex and GPVI are of particular interest because these receptors are essentially platelet specific, are critical for initiation of thrombus formation at arterial shear rates, and are implicated in wider platelet functions beyond hemostasis and thrombosis, as well as platelet aging and clearance. (Gardiner etal., 2014).

GP VI is thought to be the major signaling receptor involved in platelet activation on exposed collagen. Following GP VI interactions with collagen, platelets initiate strong activation and release the content of alpha and dense granules.( Yun etal.,2016) GPVI expression was upregulated in megakaryocytes after TPO stimulation (Holmes etal., 2002). Eltrombopag could upregulate GPVI expression in ITP patients, thereby enhancing their platelet adhesion capacity leading to reduce bleeding symptoms (Chiou etal.,2015).

The Aim is to :

To investigate the efficacy, & the safety and tolerability of eltrombopag therapy for children with persistent and chronic immune thrombocytopenia as well as the ability of eltrombopag to enhance the platelet activation through the up-regulation of glycoprotein VI (GPVI) receptor expression in comparison with other lines of treatment.

Study methods :

This study will include 40 pediatric patients with chronic or persistent ITP, age ≥ 1 to ≤ 18 years, recruited from the Hematology clinic of pediatric hospital Ain Shams University

* Baseline bleeding score assessment (ITP-BAT (v1.0) score) and Health related quality of life based on Kids' ITP Tools (KIT) questionnaires will be done.
* Patients will be divided into 2 groups:

  1. Group 1 (eltrombopag arm n=20 patients): Patients who showed no response (platelet count ≤ 20x109/L) initially for 3 months or relapse after 6 months after at least one prior ITP therapy. patients will receive a total daily dose of eltrombopag of (25-50mg/d). Dose adjustments may be made based on platelets count with an increment of 25mg once per day at 2 weeks intervals (Maximum dose: 75 mg orally once a day). If platelet counts reached more than 200 × 109 per L, the dose will be decreased by 25 mg once per day at 2 weeks intervals. If platelet counts increased to more than 400 × 109 per L, treatment will be interrupted until platelet counts decreases to less than 150 × 109 per L then the dose will be resumed at the next lower dose.

     Patients, who responded poorly to eltrombopag in 6 months or developed adverse effects, will be asked to discontinue the medication. Those who responded will be followed for further 6 month period.
  2. Group 2 (n=20 patients) Patients who are currently receiving other lines of treatment (steroids, IVIG, azathioprine, and rituximab).
* All patients will be followed clinically every 2 weeks throughout the period of the study for safety and efficacy, and complete blood counts.
* Baseline and at week 24 bone marrow examination with reticulin stain will be done
* Baseline and every 3 months liver and kidney function tests. Throughout the study periods, patients with increased serum alanine transaminase (ALT) ≥ 3 times upper limit normal (ULN) with a total bilirubin ≥2 times ULN or those with increased serum ALT ≥ 5 times ULN will be withdrawn, as well as patients with increased serum creatinine above ULN.
* Adverse events, episodes of bleeding and bleeding score will be collected and evaluated every month throughout the study.
* Health related quality of life based on Kids' ITP Tools (KIT) questionnaires will be repeated at the end of study period.
* Assessment of soluble form of glycoprotein VI using sandwich enzyme-linked immunosorbent assay (ELISA) as well as assessment of platelet activation by GPVI using flowcytometry (Gardiner, etal.,2010 ) at baseline and at the end of 6 months treatment period

Statistical Analysis : Analysis of data will be done using Statistical Program for Social Science version 21 (SPSS Inc., Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 1 to ≤ 18 years at enrollment. Patient should be able to swallow tablet form. Weight should be ≥ 12kg.
* Diagnosis of persistent (3-<12 months duration) or chronic cases (≥12 months duration) with day 1 platelet count ≤ 20x10^9.
* Patients have a bleeding score grade 3 for skin and/or grade 2 or higher for mucosal domains and/or higher than grade 1 for organ domain at the baseline visit or the worst bleeding incident episode in the patient's medical reports in the last 3 months prior screening, using ITP-BAT (v1.0) score.
* Normal Kidney function tests and liver function tests.

Exclusion Criteria:

* Acute thrombocytopenic purpura patients or Other causes of thrombocytopenia. Patients with Evans syndrome
* Hypertension, cardiovascular disease, diabetes, hepatitis C virus (HCV), HIV, hepatitis B surface antigen(HBsAg) seropositive status.
* Baseline bone marrow biopsy with evident fibrosis (reticulin stain grade 2 or more)
* Patients who have previously received eltrombopag.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Expression of glycoprotein VI collagen receptor | at 24 weeks
  Percentages of patients achieving increased expression of glycoprotein VI collagen receptor

SECONDARY OUTCOMES:
Complete response or response | at 24 weeks
  Percentages of patients achieving Complete response" (CR) defined as any platelet count of 100x109/L at least once throughout the study period in the absence of rescue treatment and those achieving "Response" (R) is defined as any platelet count between 50 and 100x 109/L or doubling of the baseline count at least once throughout the study period
Maintenance of response | at 24 weeks
  The maximum duration for which a patient continuously maintained a platelet count between 50 and 100x 10*9/L in the absence of rescue treatment.
Safety: Number of Patients who will have adverse events | at 24 weeks
  Number of Patients who will have adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Azza AG Tantawy, MD, Principal Investigator — Ain shams university, Faculty of medicine, Pediatric Hematology &Oncology department
Locations (1):
- Ainshams University , Faculty of medicine , Pediatric Hematology&Oncology unit, children hospital., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Still investigators did not decide about sharing individual participants data

REFERENCES:
- [Background] Mazzucconi MG, Fazi P, Bernasconi S, De Rossi G, Leone G, Gugliotta L, Vianelli N, Avvisati G, Rodeghiero F, Amendola A, Baronci C, Carbone C, Quattrin S, Fioritoni G, D'Alfonso G, Mandelli F; Gruppo Italiano Malattie EMatologiche dell'Adulto (GIMEMA) Thrombocytopenia Working Party. Therapy with high-dose dexamethasone (HD-DXM) in previously untreated patients affected by idiopathic thrombocytopenic purpura: a GIMEMA experience. Blood. 2007 Feb 15;109(4):1401-7. doi: 10.1182/blood-2005-12-015222. Epub 2006 Oct 31. PMID 17077333
- [Result] Buchanan GR. Overview of ITP treatment modalities in children. Blut. 1989 Jul;59(1):96-104. doi: 10.1007/BF00320257. PMID 2665875
- [Result] Bussel JB, de Miguel PG, Despotovic JM, Grainger JD, Sevilla J, Blanchette VS, Krishnamurti L, Connor P, David M, Boayue KB, Matthews DC, Lambert MP, Marcello LM, Iyengar M, Chan GW, Chagin KD, Theodore D, Bailey CK, Bakshi KK. Eltrombopag for the treatment of children with persistent and chronic immune thrombocytopenia (PETIT): a randomised, multicentre, placebo-controlled study. Lancet Haematol. 2015 Aug;2(8):e315-25. doi: 10.1016/S2352-3026(15)00114-3. Epub 2015 Jul 28. PMID 26688484
- [Result] Chiou TJ, Chang YF, Wang MC, Kao CW, Lin HY, Chen TY, Hsueh EJ, Lan YJ, Sung YC, Lin SF, Bai LY, Chen CG. Eltrombopag enhances platelet adhesion by upregulating the expression of glycoprotein VI in patients with chronic immune thrombocytopenic purpura. Transl Res. 2015 Dec;166(6):750-761.e4. doi: 10.1016/j.trsl.2015.09.005. Epub 2015 Sep 30. PMID 26477577
- [Result] Cines DB, Blanchette VS. Immune thrombocytopenic purpura. N Engl J Med. 2002 Mar 28;346(13):995-1008. doi: 10.1056/NEJMra010501. No abstract available. PMID 11919310
- [Result] Ehrlich LA, Kwitkowski VE, Reaman G, Ko CW, Nie L, Pazdur R, Farrell AT. U.S. Food and Drug Administration approval summary: Eltrombopag for the treatment of pediatric patients with chronic immune (idiopathic) thrombocytopenia. Pediatr Blood Cancer. 2017 Dec;64(12). doi: 10.1002/pbc.26657. Epub 2017 Jun 19. PMID 28627134
- [Result] Gardiner EE, Andrews RK. Platelet receptor expression and shedding: glycoprotein Ib-IX-V and glycoprotein VI. Transfus Med Rev. 2014 Apr;28(2):56-60. doi: 10.1016/j.tmrv.2014.03.001. Epub 2014 Mar 12. PMID 24674813
- [Result] Gardiner EE, Thom JY, Al-Tamimi M, Hughes A, Berndt MC, Andrews RK, Baker RI. Restored platelet function after romiplostim treatment in a patient with immune thrombocytopenic purpura. Br J Haematol. 2010 May;149(4):625-8. doi: 10.1111/j.1365-2141.2010.08092.x. Epub 2010 Feb 8. No abstract available. PMID 20148887
- [Result] Grainger JD, Locatelli F, Chotsampancharoen T, Donyush E, Pongtanakul B, Komvilaisak P, Sosothikul D, Drelichman G, Sirachainan N, Holzhauer S, Lebedev V, Lemons R, Pospisilova D, Ramenghi U, Bussel JB, Bakshi KK, Iyengar M, Chan GW, Chagin KD, Theodore D, Marcello LM, Bailey CK. Eltrombopag for children with chronic immune thrombocytopenia (PETIT2): a randomised, multicentre, placebo-controlled trial. Lancet. 2015 Oct 24;386(10004):1649-58. doi: 10.1016/S0140-6736(15)61107-2. Epub 2015 Jul 28. PMID 26231455
- [Result] Holmes ML, Bartle N, Eisbacher M, Chong BH. Cloning and analysis of the thrombopoietin-induced megakaryocyte-specific glycoprotein VI promoter and its regulation by GATA-1, Fli-1, and Sp1. J Biol Chem. 2002 Dec 13;277(50):48333-41. doi: 10.1074/jbc.M206127200. Epub 2002 Sep 30. PMID 12359731
- [Result] Klaassen RJ, Blanchette VS, Barnard D, Wakefield CD, Curtis C, Bradley CS, Neufeld EJ, Buchanan GR, Silva MP, Chan AK, Young NL. Validity, reliability, and responsiveness of a new measure of health-related quality of life in children with immune thrombocytopenic purpura: the Kids' ITP Tools. J Pediatr. 2007 May;150(5):510-5, 515.e1. doi: 10.1016/j.jpeds.2007.01.037. PMID 17452226
- [Result] Rodeghiero F, Michel M, Gernsheimer T, Ruggeri M, Blanchette V, Bussel JB, Cines DB, Cooper N, Godeau B, Greinacher A, Imbach P, Khellaf M, Klaassen RJ, Kuhne T, Liebman H, Mazzucconi MG, Newland A, Pabinger I, Tosetto A, Stasi R. Standardization of bleeding assessment in immune thrombocytopenia: report from the International Working Group. Blood. 2013 Apr 4;121(14):2596-606. doi: 10.1182/blood-2012-07-442392. Epub 2013 Jan 29. PMID 23361904
- [Result] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182
- [Result] Yun SH, Sim EH, Goh RY, Park JI, Han JY. Platelet Activation: The Mechanisms and Potential Biomarkers. Biomed Res Int. 2016;2016:9060143. doi: 10.1155/2016/9060143. Epub 2016 Jun 15. PMID 27403440
- [Result] Meletis J, Katsandris A, Raptis SD, Mantzourani M. Successful treatment of Immune Thrombocytopenic Purpura (ITP) with the thrombopoietin-mimetic romiplostim. Med Sci Monit. 2010 Aug;16(8):CS100-2. PMID 20671616